CLINICAL TRIAL: NCT05871658
Title: Efficacy of Electroacupuncture in NMOSD Patients With Pain: Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanqi Zhao,MD (Other)
Responsible Party: Sponsor-Investigator, Yuanqi Zhao,MD, director, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230221
Record Dates: First submitted 2023-04-20; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Pain
MeSH Terms: conditions — Neuromyelitis Optica; Pain | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: the electroacupuncture group (experimental group) and the sham electroacupuncture group (control group)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the electroacupuncture group (Experimental): electroacupuncture were inserted into bilateral Zusanli (ST36), Sanyinjiao (SP6), Hegu (LI4) and Quchi (LI11), and Yintang (EX-HN3). Electroacupuncture parameters selected the sparse wave, the frequency was 4 Hz, the stimulation intensity was tolerated by the patient.
  Interventions: Behavioral: electroacupuncture
- the sham electroacupuncture group (Sham Comparator): According to the previous trial,[19] sham acupoints were 1cm away from the level of the acupoints used in the EA group, which avoided the area corresponding to any of the 14 meridians of TCM. The insertion of the needle was shallower (less than 0.2cm) and had similar pain to that of normal needle insertion. The stimulation intensity was 0mA. However, the model of electroacupuncture, the frequency, and duration of treatment in the SEA group were identical in the TA group.
  Interventions: Behavioral: electroacupuncture

INTERVENTIONS:
Behavioral: electroacupuncture — electroacupuncture were inserted into bilateral Zusanli (ST36), Sanyinjiao (SP6), Hegu (LI4) and Quchi (LI11), and Yintang (EX-HN3). Electroacupuncture parameters selected the sparse wave, the frequency was 4 Hz, the stimulation intensity was tolerated by the patient.

SUMMARY:
Abstract Background Neuropathic pain is a common complication in neuromyelitis optica spectrum disorder (NMOSD), which seriously affects the quality of life of NMOSD patients, with no satisfactory treatment. Through the previous literature study and clinical observation, we found that acupuncture has good curative effect in the treatment of pain, especially electric acupuncture, but thestudies on acupuncture intervention in pain of NMOSD are still scare.

Objective To evaluate the clinical efficacy of electroacupuncture on NMOSD patients with pain.

Materials and Methods In this exploratory randomized controlled study, NMOSD patients with pain were recruited from March 21, 2022 to February 21, 2023. Patients meeting the inclusion and exclusion criteria were randomly assigned to the electroacupuncture group (experimental group) and the sham electroacupuncture group (control group) by simple random method (envelope method) according to the inclusion order. Totally, there are 20 patients enrolled.

The experimental group received electroacupuncture therapy and the control group received sham electroacupuncture therapy. A total of 8 sessions were given twice a week for 30 minutes each. On the baseline, demographic information, medication history, specimens of routine blood, blood biochemistry, liver function, IL - 6, TNF-α were collected, the brain, cervical and thoracic MRI were perfected and collected, patients filled in the SF - MPQ, NRS, SF - 36, SAS, SDS, EDSS. After the treatment, specimens of routine blood, blood biochemistry, liver function, IL - 6, TNF-α were collected again, patients filled in the SF - MPQ, NRS, SF - 36, SAS, SD, EDSS. The main outcome indicators were SF-MPQ, and the secondary outcome indicators were EDSS, NRS, SAS, SDS, SF-36, IL-6, and TNF-α.

Conclusion This is the first exploratory randomized controlled study to evaluate the efficacy of electroacupuncture on pain in patients with NMOSD. The study will provide clincial evidence of the practice of electroacupuncture on NMOSD with pain.

Key Words neuromyelitis optica spectrum disorders; pain; electroacupuncture

ELIGIBILITY:
Inclusion Criteria:

1. people diagnosed as NMOSD according to the International Panel for NMO Diagnosis (IPND) criteria.[21]
2. NRS≥4.
3. people were treated with stable doses of biological therapy and/or prednisone, with no regimen adjustment within 30 days prior to enrollment.
4. people did not adjust any standard pain medication combinations, including antiepileptic drugs, antidepressants, and opioids, within 30 days before enrollment.
5. people or their families provided written informed consent.

Exclusion Criteria:

1. people enrolled in other clinical studies.
2. people with low cognitive or mental ability.
3. people who became pregnant during the study period, breastfed, or planned to become pregnant.
4. people with serious diseases related to the heart, liver, kidney or hematopoietic system.
5. people with diabetic peripheral neuropathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Short-Form of McGill Pain Questionnaire(SF - MPQ) | on the baseline
  higher scores mean a worse outcome.
Short-Form of McGill Pain Questionnaire(SF - MPQ) | through study completion, an average of 1 month
  higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Expanded Disability Status Scale(EDSS) | on the baseline
  higher scores mean a worse outcome.
Expanded Disability Status Scale(EDSS) | through study completion, an average of 1 month
  higher scores mean a worse outcome.
numerical rating scale(NRS) | on the baseline
  higher scores mean a worse outcome.
numerical rating scale(NRS) | through study completion, an average of 1 month
  higher scores mean a worse outcome.
Self-Rating Anxiety Scale (SAS) | on the baseline
  higher scores mean a worse outcome.
Self-Rating Anxiety Scale (SAS) | through study completion, an average of 1 month
  higher scores mean a worse outcome.
Self-rating Depression Scale (SDS) | on the baseline
  higher scores mean a worse outcome.
Self-rating Depression Scale (SDS) | through study completion, an average of 1 month
  higher scores mean a worse outcome.
36-item Short-Form (SF-36) | on the baseline
  higher scores mean a better outcome.
36-item Short-Form (SF-36) | through study completion, an average of 1 month
  higher scores mean a better outcome.
Interleukin-6 (IL-6) | on the baseline
  higher scores mean a worse outcome.
Interleukin-6 (IL-6) | through study completion, an average of 1 month
  higher scores mean a worse outcome.
tumor necrosis factor-α （TNF-α） | on the baseline
  higher scores mean a worse outcome.
tumor necrosis factor-α （TNF-α） | through study completion, an average of 1 month
  higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao yuan qi, Dr, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05871658/Prot_000.pdf
  • Informed Consent Form (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05871658/ICF_001.pdf